CLINICAL TRIAL: NCT05835492
Title: A Pragmatic Real-world Multicentre Observational Research Study to Explore the Clinical and Health Economic Impact of myCOPD
Acronym: PROPEL myCOPD
Status: Active, not recruiting | Type: Observational
Sponsor: my mhealth Ltd (Industry)
Collaborators: North Bristol NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Cornwall Partnership NHS Foundation Trust (Network); University of Southampton (Other); West of England Academic Health Science Network (Unknown); Unity Insights Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: MMH-R05
Record Dates: First submitted 2023-03-27; First posted 2023-04-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Digital Health; Pulmonary Rehabilitation; Acute COPD Exacerbation; Hospital Readmission Reduction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Setting 1 - Hospital Readmission Reduction: North Bristol NHS Trust and University Hospitals Bristol and Weston NHS Foundation Trust (hospital readmissions reduction): Using myCOPD to support high risk patients with a primary focus on acute hospital admission discharge bundle following AECOPD. Patients who have been discharged from hospital following an AECOPD diagnosis and assessed in a follow-up clinic, including virtual wards, within 6 weeks can be included.
  Interventions: Device: myCOPD
- Setting 2 - Pulmonary Rehabilitation: Cornwall Partnership NHS Foundation Trust (increasing community care provision of PR): Using myCOPD to support delivery of PR and self-management in the community.
  Interventions: Device: myCOPD

INTERVENTIONS:
Device: myCOPD — myCOPD is a digital self-management application (app), that supports all elements of managing COPD by creating a supported self-help environment, and in turn reduce medical visits, and hospital admissions and re-admissions. myCOPD allows for key aspects of disease management, such as PR, to be provided remotely, based on a person's self-assessment. Furthermore, it can help people with COPD manage their condition at home, or anywhere away from a clinical setting. Successful implementation of myCOPD provides an opportunity to build capacity in primary and secondary care, and community teams where a blended approach with traditional PR and myCOPD is used. Studies have shown myCOPD is able to deliver similar improvements in symptoms and exercise tolerance compared to PR exercise-classes and helps patients admitted to hospital recover more quickly at home(5)(6). myCOPD is widely deployed across the NHS and is being used by patients in different areas of the UK.

SUMMARY:
COPD is a condition which affects over 3 million people in the UK. It causes chronic symptoms including breathlessness and cough, limitations in exercise tolerance and acute exacerbations of COPD (AECOPD) which often lead to hospital admission. Current treatment for COPD includes inhaled medication and exercise programmes called Pulmonary Rehabilitation(PR) to improve exercise tolerance and resilience to AECOPD. Currently NHS respiratory services are struggling to provide support to patients with COPD, a recent-report highlighted that 75% of people with COPD are not receiving basic care. There is an increasing need therefore to improve the provision of PR and to support patients to self-manage their condition effectively, this requires new approaches and pathways of care. My mhealth Limited MMH is a UK based digital healthcare company established in 2011, specialising in the development of digital solutions for the management of long-term conditions. Evidence based, UKCA classified, and highly secure the company has developed a suite of solutions NHS approved and widely used, MHRA registered and is working towards NICE accreditation to manage patients with asthma, COPD, diabetes, and heart disease. myCOPD is a digital self-management application (app)therapeutic, developed by MMH, that supports all elements of managing COPD by creating a supported self-help environment, and in turn reduce medical visits, and hospital admissions and re-admissions. myCOPD allows for key aspects of disease management, such as PR, to be provided remotely, based on a person's self-assessment. Furthermore, it can help people with COPD manage their condition at home, or anywhere away from a clinical setting. Successful implementation of myCOPD provides an opportunity to build capacity in primary and secondary care, and community teams where a blended approach with traditional PR and myCOPD is used. Studies have shown myCOPD is able to deliver similar improvements in symptoms and exercise tolerance compared to PR exercise-classes and helps patients admitted to hospital recover more quickly at home. myCOPD is widely deployed across the NHS and is being used by patients in different areas of the UK- but to enable NICE approval and re-imbursement across all the NHS, evidence for the health-economic benefits of its use is required.

With funding from SBRI Phase 3 grant, this project will explore the implementation of myCOPD by NHS respiratory services in two regions with diverse populations and challenges. In Bristol (Setting 1) the investigators will assess the value of using myCOPD in the COPD discharge care bundle for patients admitted to hospital with AECOPD, and its ability to help accelerate recovery, and prevent unscheduled care visits and re-admissions. Data collected from a pilot will be used to support the analysis. Whilst in Cornwall (Setting 2) the investigators will work with local services to provide 'digitally-supported PR' to isolated communities and increase the service capacity, completion rates and access to specialist support for self-management.

A formal assessment will provide vital evidence for the value of myCOPD in the NHS and enable us to develop a business case for its national adoption and use, which will ultimately transform outcomes for people with this common and complex condition.

DETAILED DESCRIPTION:
It is estimated that COPD will become the 3rd leading cause of death worldwide by 2030. COPD is a disabling, smoking related lung disease that is associated with symptoms of shortness of breath, cough, and wheeze. The natural history is one of progressive decline, frequently punctuated by periods of rapid worsening termed acute exacerbations (AECOPD). The functional limitation experienced by individuals with COPD, their propensity to exacerbations and the high levels of psychological and physical co-morbidities place a significant burden on health and social care systems in the UK.

Hospital admissions for COPD exacerbations have declined recently from 246.7 per 100,000 population in the financial year ending 2020 to 133.5 per 100,000 population in the financial year ending 2021. Although, rates remain high in the North of England and Midlands. The reason for this decline in admissions is complex and is likely to include displacement of primary admission diagnosis due to COVID-19, less exposure to infection risk due to lockdowns, mask wearing and an increased management of care in the community instead of hospital. Nonetheless, reported estimates calculate that COPD costs the NHS £1.9 billion each year. In the UK over 130,000 people with COPD are admitted to hospital annually due to AECOPD. Admissions cluster in Winter, driving bed-pressures, impacting on the delivery of care. Once admitted, COPD patients are particularly vulnerable to further exacerbations and readmission. Over 43% are readmitted within 3 months.

COPD cannot be cured and drives excess morbidity. Current treatment for COPD includes inhaled medication and exercise programmes known as PR to improve exercise tolerance and resilience to AECOPD. Patients should be educated on the importance of taking their medication as prescribed, and attending PR to avoid AECOPD events to prevent lung function decline. The benefits of PR are widely evidenced with confirmed improvements in dyspnoea, fatigue, quality of life and exercise capacity. Despite this, the proportion of patients being referred to and completing PR remains low in the UK. Early PR after hospital discharge following AECOPD has been found to reduce the risk of hospital readmission and improve quality of life. Access to PR, an essential aspect of care, is poor in the UK and in rural areas there is little or no provision. Poor provision of PR and wide geographical variation in delivery has been highlighted. Consequently, there is a significant need to explore additional strategies to support patients and healthcare professionals (HCP) in preventing or highlighting the risk of an exacerbation event.

The reasons for PR non-attendance are multifactorial and include barriers such as work or caring commitments, lack of motivation, hospitalisation or feeling unwell, transportation, or forgetting the appointment. Since COVID-19, many healthcare services turned to digital health to support remote PR delivery in the UK. This has enabled inclusion of those who would not necessarily have attended in-person PR. Patient education is key to preventing worsening of lung function. Facilitating better access to PR and smoking services will improve quality of life and relieve the growing burden on healthcare services in the UK.

myCOPD, a digital health self-management app for patients with COPD, has been in use within the NHS since 2016. It was designed by MMH, a UK based company founded by NHS respiratory consultants and is one of four long term condition self-management apps developed by the company. All MMH apps, including myCOPD, are cloud-based, meaning data is stored, managed, and processed on a network of remote servers hosted on the internet, rather than on local servers or personal computers. The apps can be accessed using any internet connected device and by download from the Apple or Google play app store. Furthermore, myCOPD provides digital disease specific support to thousands of users through self-management plans, comprehensive education on lifestyle, device instruction (inhalers), PR, symptom, COPD Assessment Test (CAT) score and exacerbation recording, and the ability to map health trends so the user and HCPs can view health deterioration or improvement over time. Recent research studies have shown the app has many benefits for both patients and healthcare service providers including a reduction in CAT score, hospital admissions and readmissions, less frequent exacerbations and improvements in inhaler technique.

The aim of this study is to use mixed-methods to understand the impact of implementing myCOPD in the NHS in the real-world. The investigators will evaluate clinical and health economic outcomes to provide essential evidence for the development of clinical pathways and business cases to enable widespread adoption of the technology across the NHS.

The investigators will explore the impact of myCOPD in supporting patients in two distinct clinical settings where the app is currently in use:

* Setting 1: University Hospitals Bristol and Weston NHS Foundation Trust and North Bristol NHS Trust will use myCOPD to support hospital discharge following AECOPD.
* Setting 2: Cornwall Partnership NHS Foundation Trust will use myCOPD to support delivery of PR and self-management in the community.

This study will require Research Ethics Committee (REC) approval.

This is a mixed-methods prospective pragmatic real-world multicentre observational study funded through the SBRI 21 Phase 3 Grant for Respiratory Diseases, led by MMH.

The trial will explore the clinical efficacy and health economic impact of a digital COPD self-management app; myCOPD, in two secondary care settings for patients with COPD. Both settings will be supported through SBRI grant funding.

The required outcomes are to collect real-world data on the efficacy of implementing a remote self-management digital health app. The focus will be on exploring its acceptability and adherence following hospital discharge and in PR delivery, and it's health economic impact.

Digital health support teams including Digital Health Champions (DHC) and Digital Health Advisors (DHA) are in place in both settings. They help break down barriers that people face to being online, improve understanding and awareness of the internet and inspire them to make digital part of their everyday lives. They offer assistance with setting up the app, how to use it, and troubleshoot.

Quantitative In both settings, participants will be offered the myCOPD app to use as an additional COPD support tool. Study assessment data will be recorded electronically using an electronic data capture (EDC) tool, and the myCOPD app for those who have chosen to use it. Data analyses will be undertaken to observe the uptake, activation, usage and engagement of myCOPD. Demographic data will be utilised to ensure that the enrolled patient group is representative of each local COPD population, considering the potential impact on health inequalities and digital exclusion. Patient reported outcome measure including COPD Assessment Test (CAT), quality of life (EQ5D-5L), Modified Medical Research Council Dyspnoea Scale (mMRC) will be analysed during the study to determine any changes for all study participants, including the sub-group who declined to use the app. Results from the Incremental Shuttle Walk Test (ISWT) will be used to determine improvements in exercise capacity before and after pulmonary rehabilitation.

In late 2022, an evaluation funded through NHSx Transformation Funding - NHS BNSSG ICB Pilot, took place within Bristol and surrounding areas. The aim of evaluation was to assess the effectiveness of using 'Digital Health Champions' (DHCs) to enrol patients onto the myCOPD application. The evaluation specifically looked at the potential benefits in excess of those observed for myCOPD as a platform (as evidenced in recent real world feasibility trials). The outcomes of this evaluation suggested that the usage of DHCs could lead to benefits beyond the level identified in unsupported trials, suggesting that the role could be used to successfully engage patients in using the application and manage their condition. The evaluation was largely assumption-based due to the availability of outcome data. It is proposed that the longer term outcomes for this patient cohort is observed as part of this study to provide further assurance of the benefits that have been realised. Data collected will also be utilised to inform health economic analysis in the form of both cost-benefit analysis from a healthcare system perspective, as well as a budget impact model, from the perspective of a single ICS.

Qualitative Real-world piloting of the implementation resources will be conducted in healthcare teams to ensure our roll-out is as acceptable and effective as possible. As the implementation is rolled out across remaining sites, further qualitative interviews with health care professional stakeholders to understand barriers to long term use, which aspects of the implementation process worked well, where improvements could be made and any issues that might inhibit full engagement will be conducted.

The investigators will conduct 8-10 semi-structured interviews with targeted patients, healthcare professionals and key stakeholders (healthcare professionals, policymakers, commissioners, technology experts, commercial partners), focusing on likely barriers e.g. time pressures and development of professional skills, perceptions of benefit, access from rural areas. The investigators will consider this with reference to existing data from myCOPD, psychological and behavioural theories to optimise implementation and meet the needs of patients and HCPs.

ELIGIBILITY:
Inclusion Criteria:

Setting 1:

* Adult patients over 18 years of age and able to give informed consent
* A clinical diagnosis of COPD
* Admitted to hospital with a primary diagnosis of AECOPD
* Assessed in a follow-up clinic and/or virtual ward within 6 weeks of an AECOPD

Setting 2:

* Adult patients over 18 years of age and able to give informed consent
* A clinical diagnosis of COPD, deemed suitable by the local clinical team as suitable for referral for PR
* Motivated/willing to take part

Exclusion Criteria:

Setting 1:

* Under 18 years of age
* No clinical diagnosis of COPD
* End of life care/palliative care
* Unable to give informed consent

Setting 2:

* Unstable angina
* MI within 6 weeks
* Uncontrolled cardiac arrhythmias
* Unstable hypertension
* Severe cognitive impairment
* Locomotor or other severe medical conditions
* Unable to give informed consent
* Any condition deemed by the PI to make the participant unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Setting 1: Participants with a COPD diagnosis who have been admitted to hospital following an acute exacerbation of COPD
  Setting 2: Participants with a COPD diagnosis who have been referred for pulmonary rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Setting 1 - Hospital Readmission Reduction | At Baseline, Months 2, 3, 6, 9, 12
  myCOPD could support patients to self-manage at home with clinical oversight by reducing the risk of hospital readmission as part of the respiratory discharge bundle. Outcome will be measured by mean change in the number of reported COPD exacerbations over 12 months. Healthcare resource utilisation over 12 months including primary care using Electronic Health Record data where possible. Data relating to each patient's admissions during the 12 months prior to enrolment will also be collected. Improved patient welfare and quality of life. Mean change in results at the end of the data collection window, compared to baseline, will be aggregated and measured against the counterfactual.
Setting 2 -Pulmonary Rehabilitation Uptake, Delivery and Completion | 12 months
  Using a digital blended approach could improve PR delivery. This outcome will be measured using the percentage of PR course completion i.e., how many sessions were attended during the 6 weeks of PR including (6 F2F sessions, 6 telephone sessions) and % of attendance. App PR course access will also be included.
Qualitative Interviews | 12 months
  Addressing potential impacts of digital-exclusion and inequality-of-access. Semi-structured interviews with targeted patients, healthcare professionals and key stakeholders (e.g. policymakers, commissioners, technology experts, commercial partners), focusing on likely barriers e.g. time pressures, perceptions of usefulness, perceived digital literacy will be conducted.

SECONDARY OUTCOMES:
Mean change in COPD Assessment Test | At Baseline, Months 2, 3, 6, 9, 12
  This is a validated symptom scoring system used in COPD studies The CAT questionnaire contains eight questions and provides a reliable measure of the impact of COPD on health status. Patients read the two statements for each item, which describe the best and worst scenario, (e.g I never cough - I cough all the time), and decide where on the scale of 0-5 they fit. The maximum score is out of 40. The higher the CAT score the greater the impact of symptoms on their health status. Experts involved in the development of CAT suggest that any change of 2 or more in the patient's final score may indicate a clinically significant change. CAT will be recorded at the start prior to any intervention at visit one, at monthly telephone calls for the duration of the study and at end of study visit
Mean change in Quality of Life Ratings measured using EuroQol 5D-5L | At Baseline, Months 2, 3, 6, 9, 12
  The EQ5D 5L is a validated questionnaire which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Minimum score is 5 and maximum score is 25 patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' score maximum 100 and 'The worst health you can imagine score minimum 0.
Mean change in Modified Medical Research Council Dyspnoea Scale | At Baseline, Months 2, 3, 6, 9, 12
  The mMRC is used to assess the degree of baseline functional disability due to dyspnoea (breathlessness). The scale measures perceived respiratory disability, using the World Health Organization (WHO) definition of disability being "any restriction or lack of ability to perform an activity in the manner or within the range considered normal for a human being".
Health Economic Analysis | 12 months
  A Cost-Benefit Analysis will capture the impact upon healthcare services through attendances and prescriptions avoided, and the impact upon patients through Quality of Life improvements (EQ-5D-5L). Primary benefit streams are expected to be reduction in readmissions, reduction in Primary Care attendances, reduction in inhaler waste and quality of life improvement. Further benefits my be incorporated into the model. Each benefit will be valued using the latest available cost data from real-world sources. Evidence will be assessed for potential uncertainty, with an appropriate Optimism Bias applied to ensure that the final model is prudent and reasonable. Outcomes will be presented in the form of a benefit-cost ratio and total cost-benefits per year at Net Present Value (NPV). This will include environmental social benefit, such as reduced carbon expenditure in attending clinical services in terms of travel saved.
Incremental Shuttle Walk Test | Baseline, month 2
  Setting 2 only, the ISWT is a symptom-limited, externally paced test, conducted along a 10 m course. The walking speed increases every minute until the patient is too breathless or fatigued to continue or can no longer maintain the required speed. The result is presented as the total distance achieved. It is reproducible after a single practice test. The change in the distance walked in the ISWT can be used to evaluate the effectiveness of an exercise training program and / or to track the change in exercise capacity over time. The minimal important difference in the distance walked is an improvement of 35m
Unscheduled Healthcare Use | At Baseline, Months 2, 3, 6, 9, 12
  Healthcare usage will apply to any participant interaction with a health care professional which involves their COPD care. This includes any interaction with GPs, practice nurses, Community, tertiary services, virtual wards, pulmonary rehabilitation programmes, radiology or other investigations associated with their COPD. Data to be recorded will be the date of interaction, reason, by whom, and whether the event was a COPD exacerbation.
myCOPD App Use | Months 6, 12
  App usage analysis measures how many features of the application patients accessed, and how consistently they were used, to support an understanding of how successfully patients engaged with the platform. This is unlikely to have a direct impact upon the listed endpoints but will provide important context in terms of the utility of the platform and which cohorts may be more or less likely to engage with them. The myCOPD clinician dashboard enables the healthcare teams to review patient reported data and app activity. Using this for monitoring patients could support the development of clinical pathways.
myCOPD App Feedback | End of Study (12 months)
  The my mhealth feedback questionnaire is based on the NHS Friends and Family Test (FFT) guidelines. This is an important feedback tool that supports the fundamental principle that people who use health services should have the opportunity to provide feedback on their experience. This is a short questionnaire consisting of multiple choice and semi structured questions. No scale is in place for this questionnaire. They will be provided to both patients and clinicians using myCOPD.
Digital Accessibility and Support | At Baseline, Months 2, 3, 6, 9, 12
  For participants who choose to use the myCOPD app, a Digital Health Advisor and/or Digital Health Champion, and/or equivalent will routinely contact the user to provide technical support with using the app. The number of times each participant has required this support will be recorded.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Cornwall Partnership NHS Foundation Trust - Liskeard Community Hospital, Liskeard, Cornwall
  - North Bristol NHS Trust - Southmead Hospital, Bristol
  - University Hospital Bristol & Weston NHS Foundation Trust - Bristol Royal Infirmary, Bristol

IPD SHARING:
Plan to Share IPD: Undecided
All results will be published in a relevant academic peer reviewed medical journal.

REFERENCES:
- [Background] National Institute for Health and Care Excellence (NICE). Chronic obstructive pulmonary disease in adults: Quality standard. NICE Guidel [Internet]. 2016;(July 2011):1-46. Available from: www.nice.org.uk/guidance/qs10/resources/chronic-obstructive-pulmonary-disease-in-adults-pdf-2098478592709
- [Background] Bollmeier SG, Hartmann AP. Management of chronic obstructive pulmonary disease: A review focusing on exacerbations. Am J Health Syst Pharm. 2020 Feb 7;77(4):259-268. doi: 10.1093/ajhp/zxz306. PMID 31930287
- [Background] Global Initiative for Chronic Obstructive Lung Disease. GOLD Report 2020. Glob Initiat Chronic Obstr Lung Dis [Internet]. 2020;141. Available from: https://goldcopd.org/wp-content/uploads/2019/12/GOLD-2020-FINAL-ver1.2-03Dec19_WMV.pdf
- [Background] Gottlieb V, Lyngso AM, Nybo B, Frolich A, Backer V. Pulmonary rehabilitation for moderate COPD (GOLD 2)--does it have an effect? COPD. 2011 Oct;8(5):380-6. doi: 10.3109/15412555.2011.610393. PMID 21936683
- [Background] Bourne S, DeVos R, North M, Chauhan A, Green B, Brown T, Cornelius V, Wilkinson T. Online versus face-to-face pulmonary rehabilitation for patients with chronic obstructive pulmonary disease: randomised controlled trial. BMJ Open. 2017 Jul 17;7(7):e014580. doi: 10.1136/bmjopen-2016-014580. PMID 28716786
- [Background] North M, Bourne S, Green B, Chauhan AJ, Brown T, Winter J, Jones T, Neville D, Blythin A, Watson A, Johnson M, Culliford D, Elkes J, Cornelius V, Wilkinson TMA. A randomised controlled feasibility trial of E-health application supported care vs usual care after exacerbation of COPD: the RESCUE trial. NPJ Digit Med. 2020 Oct 30;3:145. doi: 10.1038/s41746-020-00347-7. eCollection 2020. PMID 33145441
- [Background] World Health Organisation. Chronic Obstructive Pulmonary Disease (COPD) [Internet]. World Health Organisation. 2022 [cited 2022 Jul 14]. Available from: https://www.who.int/news-room/fact-sheets/detail/chronic-obstructive-pulmonary-disease-(copd)
- [Background] GOV.UK. Official Statistics Interactive Health Atlas of Lung conditions in England (INHALE): February 2022 update [Internet]. London; 2022. Available from: https://www.gov.uk/government/statistics/interactive-health-atlas-of-lung-conditions-in-england-inhale-2022-update/interactive-health-atlas-of-lung-conditions-in-england-inhale-february-2022-update
- [Background] The Lancet. UK COPD treatment: failing to progress. Lancet. 2018 Apr 21;391(10130):1550. doi: 10.1016/S0140-6736(18)30904-8. No abstract available. PMID 29695330
- [Background] NACAP. Drawing breath [Internet]. 2023. Available from: https://www.rcplondon.ac.uk/projects/outputs/drawing-breath-clinical-audit-report-202122
- [Background] Stone PW, Hickman K, Steiner MC, Roberts CM, Quint JK, Singh SJ. Predictors of pulmonary rehabilitation completion in the UK. ERJ Open Res. 2021 Feb 8;7(1):00509-2020. doi: 10.1183/23120541.00509-2020. eCollection 2021 Jan. PMID 33585658
- [Background] Kjaergaard J, Juhl CB, Lange P, Wilcke T. Adherence to early pulmonary rehabilitation after COPD exacerbation and risk of hospital readmission: a secondary analysis of the COPD-EXA-REHAB study. BMJ Open Respir Res. 2020 Aug;7(1):e000582. doi: 10.1136/bmjresp-2020-000582. PMID 32816829
- [Background] British Lung Foundation. Failing on the Fundamentals [Internet]. 2021. Available from: https://www.blf.org.uk/copd-report
- [Background] Sahin H, Naz I. Why are COPD patients unable to complete the outpatient pulmonary rehabilitation program? Chron Respir Dis. 2018 Nov;15(4):411-418. doi: 10.1177/1479972318767206. Epub 2018 Apr 19. PMID 29673263
- [Background] Mitchell AJ, Selmes T. Why don't patients attend their appointments? Maintaining engagement with psychiatric services. Adv Psychiatr Treat. 2007;13(6):423-34.
- [Background] Crooks MG, Elkes J, Storrar W, Roy K, North M, Blythin A, Watson A, Cornelius V, Wilkinson TMA. Evidence generation for the clinical impact of myCOPD in patients with mild, moderate and newly diagnosed COPD: a randomised controlled trial. ERJ Open Res. 2020 Oct 26;6(4):00460-2020. doi: 10.1183/23120541.00460-2020. eCollection 2020 Oct. PMID 33263052
- [Background] Kong CW, Wilkinson TMA. Predicting and preventing hospital readmission for exacerbations of COPD. ERJ Open Res. 2020 May 11;6(2):00325-2019. doi: 10.1183/23120541.00325-2019. eCollection 2020 Apr. PMID 32420313
- [Background] GOV.UK. Respiratory Disease: Applying All Our Health [Internet]. Public Health England. 2021. Available from: https://www.gov.uk/government/publications/respiratory-disease-applying-all-our-health/respiratory-disease-applying-all-our-health
- [Background] British Thoracic Society. British Thoracic Society Quality Standards for Pulmonary Rehabilitation in Adults. Br Thorac Soc Reports [Internet]. 2014;6(2). Available from: https://www.brit-thoracic.org.uk/guidelines
- [Background] Evans RA, Singh SJ. Minimum important difference of the incremental shuttle walk test distance in patients with COPD. Thorax. 2019 Oct;74(10):994-995. doi: 10.1136/thoraxjnl-2018-212725. Epub 2019 May 30. PMID 31147399